CLINICAL TRIAL: NCT04767217
Title: Evaluation of the Efficacy of Artemether-lumefantrine and Dihydroartemisinin-piperaquine in Children With Uncomplicated Clinical Malaria in Rural Rwanda
Brief Title: Malaria Therapeutic Efficacy Study, Rwanda
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Ministry of Health, Rwanda (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014153
Record Dates: First submitted 2021-02-11; First posted 2021-02-23 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Uncomplicated Malaria
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artemether-lumefantrine (ALN) (Active Comparator)
  Interventions: Drug: artemether-lumefantrine (ALN)
- dihydroartemisinin-piperaquine (DHA-PPQ) (Active Comparator)
  Interventions: Drug: dihydroartemisinin-piperaquine (DHA-PPQ)

INTERVENTIONS:
Drug: artemether-lumefantrine (ALN) — Assessing the efficacy on current 1st line antimalarial, and an alternative 1st line or 2nd line medicine
  Arms: artemether-lumefantrine (ALN)
Drug: dihydroartemisinin-piperaquine (DHA-PPQ) — dihydroartemisinin-piperaquine (DHA-PPQ)
  Arms: dihydroartemisinin-piperaquine (DHA-PPQ)

SUMMARY:
WHO recommends that Therapeutic Efficacy Studies (TES) for 1st and 2nd line antimalarial medicines should be routinely carried out and data made available for decision-making due to the threat of emergence and spread of artemisinin resistance in malaria-endemic countries, especially in Africa. In line with this WHO recommendation, Rwanda Ministry of Health (MOH) is conducting the TES to determine the efficacy of artemether-lumefantrine (ALN), which has been used in Rwanda for the last 14 years) and dihydroartemisinin-piperaquine (DHA-PPQ), another WHO-approved drug for the treatment of uncomplicated malaria which, though, has not been used in Rwanda, is being considered for adoption as a second line or alternative first line treatment. The objective of this study is to inform the decisions or actions made by a public health authority (Rwanda Rwanda Ministry of Health) to inform decision on revision of the antimalarial guidelines and policy in Rwanda. Jhpiego's Impact Malaria project in Rwanda, with funding and technical oversight from US President's Malaria Initiative (PMI) through USAID and CDC, will support the Rwanda MOH in its effort to evaluate the efficacy of ALN and DHA-PPQ in the treatment of children with uncomplicated malaria. The study is being conducted by Rwanda MOH, with technical support and funding by PMI-USAID through Jhpiego in Rwanda.

DETAILED DESCRIPTION:
WHO recommends that Therapeutic Efficacy Studies (TES) for 1st and 2nd line antimalarial medicines should be routinely carried out and data made available for decision-making due to the threat of emergence and spread of artemisinin resistance in malaria-endemic countries, especially in Africa. The Rwandan Ministry of Health (MOH) in 2006 adopted WHO-approved artemether-lumefantrine (ALN) as the first-line drug for the treatment of uncomplicated Plasmodium falciparum malaria. A clinical trial carried out in 2004-2005 in Rwanda showed that ALN was very efficacious in children although efficacy varied in different parts of the country. ALN efficacy was shown to remain high in TES conducted in 2012-2015 and in 2018. However, both studies found a molecular marker of parasite resistance to artemisinin (included delayed parasite clearance associated with artemisinin resistance in one site in 2018) and both studies also found high prevalence of markers associated with tolerance to lumefantrine. The clinical efficacy of ALN therefore needs to be regularly monitored in Rwanda to ensure this first line treatment is still efficacious. Given the detection of antimalarial resistance markers in recent TES, it is also important for Rwanda MOH to determine the efficacy an additional ACT that could be considered for adoption as a second line or alternative first line treatment. This study will monitor the efficacy of ALN (which has been used in Rwanda for the last 14 years) and dihydroartemisinin-piperaquine (DHA-PPQ), another WHO-approved ACT for the treatment of uncomplicated malaria which has not been used in Rwanda.

In line with the WHO recommendation, Jhpiego Impact Malaria project in Rwanda, with funding and technical oversight from US President's Malaria Initiative (PMI) through USAID and CDC, will be supporting the Rwanda MOH Malaria and Other Parasitic Diseases Unit (MOPDD) of the Rwanda Biomedical Center (RBC) to conduct a TES to monitor the efficacy of ALN and DHA-PPQ in children with uncomplicated clinical malaria in rural Rwanda. The study is being conducted by Rwanda MOH MOPDD, with technical support and funding by PMI-USAID through the Jhpiego Impact Malaria project in Rwanda.

Objective: To evaluate the efficacy of artemether-lumefantrine (ALN) and dihydroartemisinin-piperaquine (DHA-PPQ) in children with uncomplicated clinical malaria in rural Rwanda

Study Sites: The study will be conducted in three sentinel sites - Rukara, Bugarama and Masaka rural health centers- where antimalaria efficacy studies are always carried out in Rwanda because of the intensity of malaria transmission. Different levels of artemisinin resistance have been identified in two of these three (Rukara and Bugarama) in previous studies. At each site, there will be two arms: one for ALN and one for DHA-PPQ.

Study Design: The study will be a two-arm, open-label trial in which patients (children aged 6 months to 59 months) with uncomplicated P. falciparum malaria will be treated with supervised doses of ALN or DHA-PPQ. Children will be followed for 28 days after treatment for ALN and 42 days after DHA-PPQ. Data on molecular markers of artemisinin resistance will be collected at all sites. The study will be conducted at three sites in Rwanda with historically different efficacy profiles to antimalarials, including ACTs.

The primary endpoint is the clinical and parasitological cure by day 28 (ALN) and day 42 (DHA-PPQ) post-treatment.

Study Period: March 2021 to October 2022

Sample Size: At each site, 88 patients per treatment arm (allowing for 20% loss to follow-up) would be enrolled. In total, we will enrol 528 patients in our study.

Treatment(s) and follow-up: All children enrolled in the study will be admitted to a health centre for three days to ensure adherence to treatment regimen, and detect possible adverse events. Clinical and parasitological parameters will be monitored over a 28-day follow-up period to evaluate ALN efficacy, and over a 42-day follow-up period to evaluate DHA-PPQ efficacy.

Exploratory endpoints: to characterize molecular markers of artemisinin and partner drug resistance in all three sites and the clinical (parasite clearance) and in vitro phenotypes of resistance in two of the three study sites: Rukara and Masaka.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 59 months old
* Monoinfection with P. falciparum and parasitaemia of 1,000 - 100,000 asexual parasites per µl
* Axillary temperature 37.5 °C or history of fever in the preceding 24 hours before recruitment
* Ability to swallow oral medication
* Haemoglobin ≥7.0 g/dL at admission
* Informed consent from guardian/parent of patient
* Parent/guardian agrees to bring the patient for planned follow-up visits at day 7, 14, 21, 28, 35, and 42 (35 and 42 in DHA-PPQ arm only)
* Ability for the child to be admitted to a health center for inpatient blood testing, observation and treatment for three days

Exclusion Criteria:

* Danger signs of severe malaria or signs of severe malaria
* Other underlying diseases (cardiac, renal, hepatic diseases)
* Severe malnutrition according to WHO child growth standards (WHO, 2006), children - with marasmus or oedematous malnutrition
* History of allergy to study drugs
* A clear history of receiving any antimalarial treatment in the preceding 72 hours
* Ongoing prophylaxis with drugs having antimalarial activity, such as cotrimoxazole for the prevention of Pneumocisti jirovici pneumonia in children born to HIV+ women

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 528 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Number of patients (in the artemether-lumefantrine arm) with clinical and parasitological cure (i.e. free of malaria symptoms and parasites) assessed clinically and via microscopy and rapid diagnostic test | By day 28 post-treatment
Number of patients (in the dihydroartemisinin-piperaquine arm) with clinical and parasitological cure (i.e. free of malaria symptoms and parasites) assessed clinically and via microscopy and rapid diagnostic test | By day 42 post-treatment

SECONDARY OUTCOMES:
Number of patients (in the artemether-lumefantrine arm) that developed molecular markers of drug (artemisinin) resistance (assessed via phenotype tests) | By day 28 post-treatment
Number of patients (in the dihydroartemisinin-piperaquine arm) that developed molecular markers of drug (artemisinin) resistance (assessed via phenotype tests) | By day 42 post-treatment

CONTACTS AND LOCATIONS:
Locations (3):
- Rwanda (3):
  - Bugarama health center, Bugarama
  - Masaka health center, Masaka
  - Rukara health center, Rukara

IPD SHARING:
Plan to Share IPD: No